CLINICAL TRIAL: NCT03364348
Title: A Phase 1B Dose Escalation Trial of Human Anti 4 1BB Agonistic Antibody Utomilumab (PF 05082566) in Combination With Ado Trastuzumab Emtansine or Trastuzumab in Patients With HER2 Postive Advanced Breast Cancer
Brief Title: 4-1BB Agonist Monoclonal Antibody PF-05082566 With Trastuzumab Emtansine or Trastuzumab in Treating Patients With Advanced HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: George W. Sledge Jr. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, George W. Sledge Jr., Principal Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-37299; NCI-2016-01881 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRS0070 (Other: OnCore)
Record Dates: First submitted 2017-11-10; First posted 2017-12-06 (Actual); Results first posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-09

CONDITIONS: HER2 Positive Breast Carcinoma; Recurrent Breast Carcinoma; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — utomilumab; Trastuzumab; PF-05280014; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1A (trastuzumab + utomilumab) (Experimental): Utomilumab 20 mg IV + trastuzumab 6 mg/kg IV every 3 weeks. 3 subjects will be treated at this dose level. If no DLT events are recorded, then utomilumab dose will be increased to 100 mg (Dose Level 1B).
  Interventions: Drug: Utomilumab; Drug: Trastuzumab
- Cohort 1B (trastuzumab + utomilumab) (Experimental): Utomilumab 100 mg IV + trastuzumab 6 mg/kg IV every 3 weeks.
  Interventions: Drug: Utomilumab; Drug: Trastuzumab
- Cohort 2A (ado-trastuzumab emtansine + utomilumab) (Experimental): Utomilumab 20 mg IV + ado-trastuzumab emtansine 3.6 mg/kg IV every 3 weeks.
  Interventions: Drug: Utomilumab; Drug: Ado-Trastuzumab Emtansine
- Cohort 2B (ado-trastuzumab emtansine + utomilumab) (Experimental): Utomilumab 100 mg IV + ado-trastuzumab emtansine 3.6 mg/kg IV every 3 weeks.
  Interventions: Drug: Utomilumab; Drug: Ado-Trastuzumab Emtansine

INTERVENTIONS:
Drug: Utomilumab — Given IV
  Other Names: 4-1BB Agonist Monoclonal Antibody PF-05082566; PF-05082566; PF-2566
Drug: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar PF-05280014
  Arms: Cohort 1A (trastuzumab + utomilumab); Cohort 1B (trastuzumab + utomilumab)
Drug: Ado-Trastuzumab Emtansine — Given IV
  Other Names: Trastuzumab Emtansine; Kadcyla; PRO132365; RO5304020; T-DM1; Trastuzumab-DM1; Trastuzumab-MCC-DM1; Trastuzumab-MCC-DM1 Antibody-Drug Conjugate; Trastuzumab-MCC-DM1 Immunoconjugate
  Arms: Cohort 2A (ado-trastuzumab emtansine + utomilumab); Cohort 2B (ado-trastuzumab emtansine + utomilumab)

SUMMARY:
This trial studies the best dose and side effects of utomilumab (4-1BB agonist monoclonal antibody PF-05082566) with trastuzumab emtansine or trastuzumab in treating patients with HER2-positive breast cancer that has spread to other places in the body. Monoclonal antibodies, such as utomilumab, trastuzumab emtansine, and trastuzumab may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Estimate the maximum tolerated dose (MTD) and determine the recommended dose (RP2D) of utomilumab in combination with ado-rastuzumab emtansine (T-DM1) or trastuzumab in subjects with HER2-positive advanced breast cancer.

SECONDARY OBJECTIVES:

* Determine the objective tumor response (ORR)
* Determine the time to tumor response (TTR)
* Determine the duration of response (DR)
* Determine progression free survival (PFS)
* Assess the safety and tolerability of utomilumab in combination with ado-trastuzumab emtansine or trastuzumab

OUTLINE: Patients are randomized to 1 of 2 cohorts.

COHORT 1: Dose 1: Utomilumab 20 mg IV + ado-trastuzumab emtansine (T-DM1) 3.6 mg/kg IV every 3 weeks. Dose 2: Dose Level 2 - Utomilumab 100 mg IV + ado-trastuzumab emtansine 3.6 mg/kg IV every 3 weeks

COHORT 2: Dose 1: Utomilumab 20 mg IV + trastuzumab 6 mg/kg IV every 3 weeks. Dose Level 2 - Utomilumab 100 mg IV + trastuzumab 6 mg/kg IV every 3 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

* History of biopsy proven HER2 overexpressing breast cancer and radiographic evidence of metastatic disease, or locally recurrent unresectable disease. The HER2 status can be determined either by immunohistochemistry (IHC) [IHC score, 3+] or by fluorescence in situ hybridization (FISH) [as defined by HER2/CEP 17 ratio ≥ 2.0, or HER2 copy number ≥ 6], or as otherwise defined by 2018 ASCO/CAP guidelines.
* Cohort 1 subjects must have received trastuzumab and a taxane separately or in combination (those who previously received ado-trastuzumab emtansine may accrue to Cohort 2).
* Subjects in Cohort 2 must have received at least 1 prior therapy including ado-trastuzumab emtansine.
* Subjects who discontinued prior trastuzumab or ado trastuzumab emtansine due to progressive or refractory disease are eligible for enrollment
* Available tumor samples. For eligibility, if no unstained slides remain, stained pathology slides may be reviewed at the treating institution. However, a tumor sample is required for research evaluations per the following (any of Item 1; 2; or 3, in order of preference).
* A FFPE tumor tissue block from a de novo fresh tumor biopsy obtained during screening will be requested, though not mandated.
* A recently obtained archival FFPE tumor tissue block (or 10 to 15 unstained slides) from a primary or metastatic tumor resection or biopsy if the following criteria are met:
* The biopsy or resection was performed within 1 year of enrollment OR
* The subject has not received any intervening systemic anti cancer treatment from the time the tissue was obtained and enrolled onto the current study. OR
* Any archival FFPE tumor tissue block (or unstained slides) from primary tumor resection specimen (if not provided per above). The archival sample may have been collected at any time prior to the current study, regardless of any intervening therapy. If an FFPE tissue block cannot be provided, a minimum of 10 unstained slides (15 preferable) will be acceptable.
* Subjects must have evaluable OR measurable disease, as defined by RECIST v1.1.
* Performance status 0 to 1 (by Eastern Cooperative Oncology Group [ECOG] scale).
* Laboratory parameters (must satisfy all): Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (≥ 1500/µL) Platelet count ≥ 100 × 109/L (≥ 100,000 /µL) Hemoglobin ≥ 9.0 g/dL; subjects on therapeutic anticoagulation are eligible if there is no bleeding and they are on a stable dose of anticoagulation therapy (eg, on Coumadin with an INR of 2 to 3) for at least 7 days before registration (prior to the start of therapy, or stable heparin or Factor Xa inhibitor dose) Serum creatinine ≤ 1.5 × the ULN or calculated creatinine clearance (by Cockcroft Gault formula) ≥ 60 mL/min Aspartate aminotransferase (AST) ≤ 2.5 × ULN Alanine aminotransferase (ALT) ≤ 2.5 × ULN Bilirubin ≤ 1.5 × ULN
* Subjects must not be pregnant or breastfeeding. A pregnancy test will be obtained if the subject is a woman of child bearing potential, defined as a sexually mature woman who has not undergone a hysterectomy or and/or bilateral oophorectomy or who has not been naturally postmenopausal for at least 24 consecutive months (ie, who has had menses at any time in the preceding 24 consecutive months) with 2 pregnancy tests, one at screening, and another immediately preceding the initiation of treatment.
* Subjects must have signed an informed consent document stating that they understand the investigational nature of the proposed treatment
* Left ventricular ejection fraction determined by echocardiogram or multiple gated acquisition scan (MUGA) (cardiac scan) must be 50% or higher.

EXCLUSION CRITERIA:

* Previously discontinued either trastuzumab or ado trastuzumab emtansine due to intolerance.
* Received any other investigational agents within 30 days of registration.
* Central nervous system (CNS) metastases, unless previously treated by either radiation therapy and/or surgical resection, clinically stable for at least 60 days and on a stable corticosteroid dose of ≤ 4 mg/day decadron (or equivalent steroid regimen) for at least 1 month. Subjects with a history of CNS metastases that are both treated and stably controlled are eligible if all of the following apply:
* Therapy has been administered (surgery and/or radiation therapy);
* There is no additional treatment planned for brain metastases;
* The subject is clinically stable;
* The subject is on a stable corticosteroid dose of ≤ 4 mg/day decadron (or equivalent steroid regimen) for at least 1 month.
* Prior malignancy (other than in situ cervical cancer, or basal cell or squamous cell carcinoma of the skin), unless treated with curative intent and without evidence of disease for 3 years or longer
* Administration of other prior anticancer therapies within 4 weeks of enrollment, except ongoing administration of a bisphosphonate drug or denosumab as treatment for bone metastasis
* Toxicities related to prior anticancer treatment (except alopecia) that have not resolved to ≤ Grade 1 according to common terminology criteria for adverse events (CTCAE v5) before registration or prior to start of therapy
* Currently receiving systemic antibiotic, antiviral, or antifungal therapy for the treatment of an active infection
* Systemic corticosteroid therapy at doses of greater than prednisone 5 mg daily (or dose-equivalent chronic steroid regimen) for therapeutic and not adrenal replacement indications (maintenance steroid use for adrenal insufficiency is permitted). Acute emergency administration, topical applications, inhaled sprays, eye drops or local injections of corticosteroids are allowed.
* History of bleeding diathesis
* Any co morbid medical condition deemed by the treating or principal investigator to possibly put the subject at significant risk for toxicity.
* Subject has known sensitivity to any of the products to be administered during dosing
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of venous thromboembolism within prior 6 months.
* Subject with reproductive potential who will not agree to use, during the study and for 60 days after the last dose of utomilumab or 6 months for ado trastuzumab emtansine or trastuzumab 2 highly effective method of contraceptive such as:
* Implants
* Injectables
* Intrauterine devices (IUDs) such as copper T or Levonorgestrel releasing intrauterine system (LNG IUS)
* Sexual abstinence
* Vasectomized partner
* Condom or occlusive cap (diaphragm or cervical/vault cap) supplemented with the use of a spermicide during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Sledge, MD, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1A (Trastuzumab + Utomilumab) | Cohort 1B (Trastuzumab + Utomilumab) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
Started | 3 | 2 | 3 | 10
Completed | 3 | 2 | 3 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A (Trastuzumab + Utomilumab) | Cohort 1B (Trastuzumab + Utomilumab) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab) | Total
Number analyzed (Participants) | 3 | 2 | 3 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 9 | 15
  >=65 years | 1 | 0 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 10 | 18
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 4
  Not Hispanic or Latino | 2 | 1 | 3 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 3 | 1 | 3 | 4 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 3 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities (DLTs)
Description: Dose-limiting toxicities (DLTs) within the first 2 cycles (6 weeks) of treatment were assessed. DLTs are treatment-related adverse events defined as:
  * Neutropenia Grade (Gr) 4 >7 days
  * Febrile neutropenia, defined as absolute neutrophil count <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of ≥38 degrees C (100.4 degrees F) for >1 hour
  * Neutropenic infection ≥Gr 3
  * Thrombocytopenia ≥Gr 4, or with bleeding Gr 3
  * Non-laboratory toxicities ≥Gr 3, except nausea, vomiting, or diarrhea recovering to <Gr 2 within 48 hours.
  * Laboratory abnormalities [other than aspartate aminotransferase / alanine aminotransferase (AST/ALT)] ≥Gr 3, if:
    * Medical intervention required
    * Hospitalization required, or
    * >24 hours
  * AST & ALT Gr 4, or >3×ULN
  * Total bilirubin >2×ULN, with no elevation of alkaline phosphatase The outcome is reported as the number of DLTs observed per group, a number with dispersion.
Time Frame: 6 weeks
Measure: Number; unit: Dose-limiting toxicities (DLTs)
Arm/Group | Cohort 1A (Trastuzumab + Utomilumab) | Cohort 1B (Trastuzumab + Utomilumab) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
Number analyzed (Participants) | 3 | 2 | 3 | 10
Dose-limiting toxicities (DLTs) | 0 | 0 | 0 | 0

2. Secondary Outcome: Objective Tumor Response (ORR)
Description: Objective tumor response (ORR) per RECIST v1.1 was assessed after 4 cycles (3 months) of treatment. RECIST v1.1 was assessed on target lesions as:
  * Complete Response (CR): Complete disappearance of all lesions with the exception of nodal disease. All target lymph nodes must decrease to normal size (short axis < 10 mm).
  * Partial Response (PR): ≥ 30% decrease in the sum of diameters of all measurable lesions.
  * Progressive Disease (PD): Increase in lesion size ≥ 5 mm and ≥ 20% increase in the sum of diameters of measurable lesions.
  * Stable Disease (SD): All lesions assessed, but not CR, PR, or PD.
  Per protocol, the outcome is reported for participants in Cohort 2B (ado-trastuzumab emtansine + utomilumab) as the number of participants with the indicated clinical response, a number without dispersion.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
Number analyzed (Participants) | 10
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 1
  Progressive Disease (PD) | 5
  Stable Disease (SD) | 4

3. Secondary Outcome: Time-to-tumor Response (TTR)
Description: Time-to-tumor response (TTR) was assessed per RECIST v1.1, in participants who have at least 1 on-study tumor assessment & respond within 4 cycles (3 months). RECIST v1.1 was assessed as:
  * Complete Response (CR): Complete disappearance of target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis < 10 mm).
  * Partial Response (PR): ≥ 30% decrease in the sum of diameters of target measurable lesions.
  By definition, TTR an assessment of the tumor response, meaning a CR or a PR.
  Per protocol, the outcome is reported as the median with full range for participants in Cohort 2B (ado-trastuzumab emtansine + utomilumab) achieving a clinical response within 4 cycles (3 months).
Time Frame: 3 months
Population: Not all participants in Cohort 2B achieved a clinical response within 4 cycles (3 months).
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
Number analyzed (Participants) | 1
weeks | 12 [12 to 12]

4. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response (DoR) was assessed in participants who have 1+ on-study tumor assessment(s) and have a clinical response, through up to 5 years after treatment. RECIST v1.1 was assessed as:
  * Complete Response (CR): Complete disappearance of target lesions with the exception of nodal disease. Target nodes must decrease to normal size (short axis < 10 mm).
  * Partial Response (PR): ≥ 30% decrease in the sum of diameters of target measurable lesions.
  * Progression Disease (PD): Increase in lesion size ≥ 5 mm and ≥ 20% increase in the sum of diameters of target measurable lesions.
  * Stable Disease (SD): Target lesions assessed, but not CR, PR, or PD.
  By definition, DoR is an assessment of tumor response, meaning the participants achieved a CR or a PR.
  Per protocol, the outcome is reported as the median with full range for participants in Cohort 2B (ado-trastuzumab emtansine + utomilumab) achieving a clinical response within 5 years (260 weeks).
Time Frame: up to 260 weeks
Population: This analysis includes only those Cohort 2B participants who had a Complete Response (CR) or a Partial Response (PR).
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
Number analyzed (Participants) | 2
weeks | 54 [45 to 63]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) means the participants remained alive without disease progression (DP). DP was defined per RECIST v1.1 as an increase in lesion size ≥ 5 mm or ≥ 20% increase in the sum of diameters of target measurable lesions. The outcome is reported as the median time that participants survived without DP, with full range.
Time Frame: 128 weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort 1A (Trastuzumab + Utomilumab) | Cohort 1B (Trastuzumab + Utomilumab) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
Number analyzed (Participants) | 3 | 2 | 3 | 10
weeks | 9 [6 to 15] | 15 [12 to 17] | 45 [12 to 128] | 12 [3 to 85]

6. Secondary Outcome: Adverse Events by Severity Grade 1 to 5
Description: Adverse events while receiving treatment and within 30 days were assessed by treatment group for severity (as graded by NCI CTCAE v5). The outcome is reported by treatment group as the numbers of adverse events by treatment group, numbers without dispersion.
Time Frame: Up to 128 weeks
Measure: Number; unit: adverse events
Arm/Group | Cohort 1A (Trastuzumab + Utomilumab) | Cohort 1B (Trastuzumab + Utomilumab) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
Number analyzed (Participants) | 3 | 2 | 3 | 10
adverse events
  CTCAE Grade 1 | 4 | 10 | 71 | 121
  CTCAE Grade 2 | 11 | 4 | 17 | 39
  CTCAE Grade 3 | 5 | 0 | 3 | 9
  CTCAE Grade 4 | 0 | 0 | 0 | 1
  CTCAE Grade 5 | 0 | 0 | 0 | 0

7. Secondary Outcome: Adverse Event Relationship to Study Drugs
Description: Adverse events while receiving treatment and within 30 days were assessed by treatment group for relationship to the study treatments. The outcome is reported as the numbers of related adverse events by treatment group, numbers without dispersion.
Time Frame: Up to 128 weeks
Measure: Number; unit: adverse events
Arm/Group | Cohort 1A (Trastuzumab + Utomilumab) | Cohort 1B (Trastuzumab + Utomilumab) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
Number analyzed (Participants) | 3 | 2 | 3 | 10
adverse events
  Not related | 3 | 2 | 14 | 24
  Unlikely related | 15 | 8 | 15 | 29
  Possibly related | 1 | 4 | 46 | 70
  Probably related | 1 | 0 | 11 | 49
  Definitely related | 0 | 0 | 5 | 0

8. Other Pre Specified Outcome: Laboratory Value Abnormalities
Description: Adverse events that were laboratory value abnormalities that occurred during treatment or within 30 days, were assessed by treatment group. The outcome is reported as the number of laboratory abnormalities by treatment group that were laboratory value abnormalities (Yes) or not (No), numbers without dispersion.
Time Frame: Up to 128 weeks
Measure: Number; unit: adverse events
Arm/Group | Cohort 1A (Trastuzumab + Utomilumab) | Cohort 1B (Trastuzumab + Utomilumab) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
Number analyzed (Participants) | 3 | 2 | 3 | 10
adverse events
  Yes | 1 | 2 | 18 | 18
  no | 18 | 12 | 73 | 152

ADVERSE EVENTS:
Time Frame: 128 weeks
Arm/Group | Cohort 1A (Trastuzumab + Utomilumab) | Cohort 1B (Trastuzumab + Utomilumab) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2 | 0/3 | 2/10
Other Adverse Events (participants affected / at risk) | 2/3 | 2/2 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A (Trastuzumab + Utomilumab) (N=3) | Cohort 1B (Trastuzumab + Utomilumab) (N=2) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) (N=3) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab) (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A (Trastuzumab + Utomilumab) (N=3) | Cohort 1B (Trastuzumab + Utomilumab) (N=2) | Cohort 2A (Ado-trastuzumab Emtansine + Utomilumab) (N=3) | Cohort 2B (Ado-trastuzumab Emtansine + Utomilumab) (N=10)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (7) | 5 (15)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye disorders - Other (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (7)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 3 (10) | 6 (9)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (9) | 4 (5)
Flu-like symptoms (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (3) | 1 (1) | 1 (1) | 3 (4)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (10)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 7 (11)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 5 (10)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2) | 4 (7)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 2 (5) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT03364348/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03364348/ICF_001.pdf